CLINICAL TRIAL: NCT05336955
Title: Evaluation of Telehealth Services on Mental Health Outcomes for People With Intellectual and Developmental Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Hampshire (Other)
Collaborators: University of Florida (Other); Georgetown University (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNH-08-FY2023-2-01; UNH IRB-FY2022-232 (Other: University of New Hampshire)
Record Dates: First submitted 2022-03-24; First posted 2022-04-20 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Conditions; Developmental Disability
MeSH Terms: conditions — Developmental Disabilities | interventions — Referral and Consultation; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemental health START (Experimental): Telemental health START will deliver two components via telephonic or other communication technology (e.g., Zoom). This includes component #2 (consultation and coping skills coaching) and component #4 (service linkages, referrals, outreach, & training). START components #1 (intake and quarterly assessment) and #3 (24-hour urgent crisis response and intervention) will continue to be provided in-person.
  Interventions: Other: Intake and quarterly assessment:; Other: Consultation & coping skills coaching:; Other: 24-hour urgent crisis response and intervention:; Other: Service linkages, referrals, outreach, & training:
- In-person START (Active Comparator): In-person START will deliver all model components in-person. This is the established model.
  Interventions: Other: Intake and quarterly assessment:; Other: Consultation & coping skills coaching:; Other: 24-hour urgent crisis response and intervention:; Other: Service linkages, referrals, outreach, & training:

INTERVENTIONS:
Other: Intake and quarterly assessment: — The START Plan is designed to evaluate the mental health needs of persons with IDD and measure the capacity of the formal and natural support systems. Family caregivers, or the person primarily responsible for day-to-day care of the person, participate in a formatted interview conducted by START coordinators. The START coordinator completes the initial START Plan during intake and quarterly thereafter. Based on informant responses, an intensity rating is assigned to determine the type, frequency, and duration of services to be provided. Quarterly assessment is conducted to inform development or modification of the Cross-Systems Crisis Prevention and Intervention Plan (D.2.b.2.). Hypothesized causal pathway: Family caregiver engagement in assessment enables the START team to efficiently and effectively identify needs and socially valid solutions that strategically reduce use of emergency services and increase mental health stability.
Other: Consultation & coping skills coaching: — Mental health service consultation is provided by START clinical and medical directors in order to prevent and de-escalate crises. Coping skills coaching, provided by START coordinators, helps to determine with the person, their family, and the system of care how to promote well-being and stability. Successful coping skills for the person are incorporated into the Cross-Systems Crisis Prevention and Intervention Plan. All methods are manualized and reported to meet model fidelity. Hypothesized causal pathway: Providing consultation and coping skills coaching to youth and young adults with IDD, their families, and their system of care increases capacity for crisis prevention and stabilization, reduces emergency service use, and increases quality of care, leading to long-term stability.
Other: 24-hour urgent crisis response and intervention: — START teams have 24-hour, in-person mobile crisis intervention services. Emergency calls come from a variety of sources; clients, emergency rooms, service providers, families, and law enforcement. START provides immediate telephonic response and in-person evaluation within two hours of the initial contact. Hypothesized causal pathway: Real-time, immediate support enables the successful enactment of crisis evaluation and stabilization. This reduces severity of the crises and allows for diversion from emergency service use.
Other: Service linkages, referrals, outreach, & training: — START teams work with stakeholders to develop and maintain linkage agreements. The purpose of these agreements is to enhance the capacity of the system as a whole and develop partnerships to reduce disparities and gaps in the service array. START coordinators conduct crisis prevention-focused outreach visits with the person and/or their system of care. Examples include training during home- and school-based visits, family caregiver coaching to implement new plans or strategies, and checking in with the person to monitor their level of stability. Hypothesized causal pathway: Increased person-centered collaboration and dialogue across systems of care promotes patient perceived quality of care, the identification of more effective strategies that support their mental health needs, and results in reduced use of emergency services.

SUMMARY:
Roughly 40% of those with intellectual and developmental disabilities (IDD) have mental health needs, which is twice the national average. Nevertheless, there is dearth of evidenced-based mental health treatment for youth and young adults with IDD. The disparity in access to mental health care places those with IDD at greater risk of crisis service use. While telemental health studies demonstrate potential to enhance access to care, little of this research includes those with IDD, or crisis prevention and intervention. This project will refine and evaluate telemental health services for youth and young adults with IDD delivered within START (Systemic, Therapeutic, Assessment, Resources, and Treatment), a national, evidence-based model of crisis prevention and intervention for people with IDD. The study will begin with stakeholder feedback (service recipients, families, and providers) regarding telemental health services (Aim 1). Results will be used to refine the intervention. Our team will then compare telemental health versus in-person START services in a randomized control trial (Aim 2). To our knowledge, this will be the first trial of a telemental health crisis program for the IDD population. The final goal is to understand if outcomes vary across subpopulations (Aim 3) and to identify potential disparities. If found, the investigators will work with service users, families and providers to develop a strategy to address identified disparities in outcomes. The study will be executed by an interdisciplinary team of experts engaged with stakeholder partners. Understanding the benefits of specific telemental health methods has important implications to the design of interventions, within and outside of START. This telemental health study offers promise to address disparities in access to mental health care for people with IDD.

DETAILED DESCRIPTION:
Aim 1: Refine START (Systemic, Therapeutic, Assessment, Resources, and Treatment) telemental health practices to meet the needs of persons with IDD and mental health needs, their family caregivers, and providers.

The primary goal of Aim 1 is to identify strengths and weaknesses of telemental health START practices to inform the patient-centered intervention protocols used in Aim 2. The investigators hypothesize that our engagement approach and the qualitative methods used to design the telemental protocols will result in telemental health services that are accessible, acceptable, and inclusive in response to the diverse community of people with IDD-MH and their families.

The secondary goal of Aim 1 is to design the Person Experiences Interview Survey (PEIS), adapted from the gold-standard Family Experiences Interview Schedule (FEIS). The investigators hypothesize that our engagement approach and the qualitative methods used to design the Person Experiences Interview Survey (PEIS) will result in a self-report tool with content validity for youth and young adults with IDD and mental health service experiences as indicated by the relevance, comprehensiveness, and ease of understanding.

Aim 2: Compare the effectiveness of in-person START practices versus START telemental health using a randomized control design.

It is hypothesized that telemental health START will not be inferior to in-person START in the reduction of emergency psychiatric service use, time-to-discharge, and improvement in mental health stability and perceived quality of care. This finding will support the use of telemental health practices as a valuable alternative to in-person care.

Aim 3: Evaluate heterogeneity of treatment response by assessing differences in outcomes (emergency service diversion, perceived quality of care, and mental health stability) across diverse groups (e.g., race, ethnicity, language spoken, rural settings, level of intellectual disability).

It is hypothesized that study outcomes (emergency service use, quality of care, and mental health stability) will not be inferior for the telemental health condition compared to the in- person condition within or across diverse groups, except for those living in rural settings. The investigators hypothesize improved outcomes will be found among those in the telemental health condition who live in a rural setting, compared to those living in a rural setting who are in the in-person condition, given the known difficulty in accessing in-person services for those living far from care. This finding will support equitable effects of telemental health START practices among diverse racial/ethnic and developmental groups, with potential added value for those living in rural settings.

ELIGIBILITY:
Inclusion criteria:

* participant age 12-45 years
* Lives in family setting
* New START enrollee (within 90 days of enrollment)
* Enrolled at an eligible START site
* Able to obtain informed consent.

Exclusion:

* None

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Family Experiences Interview Schedule (FEIS) over 1 year | Change in FEIS scores [at 2 timepoints: enrollment, and 1 year (or discharge)]
  A semi-structured interview of caregiver experiences with the mental health system

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) at 1 year | Change in ABC scores [at 3 timepoints: enrollment, 6 months, and 1 year (or discharge)]
  Mental health symptom checklist
Change in Crisis Service Use at 1 year | Change between enrollment to 1 year (or discharge)
  Number (and outcomes) fo contacts with the START. This outcome is continuously monitored.
Time to discharge | continuous monitoring up to 1 year
  Number of days enrolled up to 1 year
Change in mental health stability as measured by START Plan scores at 1 year | Change in START plan scores [at 3 timepoints: enrollment, 6 months, and 1 year (or discharge)
  The START Plan is a custom measure developed by and for the START project. It is a multi-informant measure of mental health and service stability. It is conducted by the START coordinator using their observations and input from primary caregivers or appropriate professional staff. Specifically, it has three sections. Section A is a historical report of mental health challenges. Section B is the level of intensity and risk of mental health challenge. Section C assesses quality of perceived professional and community supports, from both the coordinator and informant perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Beasley, PhD, Principal Investigator — University of New Hampshire
Locations (1):
- NC West, Concord, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The full data package will be maintained and made publicly available for at least 7 years. Individual Participant data (IPD) will be made publicly available after full de-identification. It will be included in the full data package. The full data package includes the de-identified IPD, full study protocol, data handbook, data dictionary, full statistical analysis plan (including all amendments and all documentation for additional work processes), and analytic code. Analytic code will be written in STATA 15.0 (College Station, Tx). Dr. Kalb (Co-PI) will serve as the contact for third party use. The full data package will be shared via PCORI's designated registry.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 7 years post study
Access Criteria: none. The full data package, including the IPD, will be made publicly available in the PCORI registry, as listed below.
URL: https://www.icpsr.umich.edu/web/pages/pcodr/

REFERENCES:
- [Background] Kalb LG, Beasley JB, Caoili A, McLaren JL, Barnhill J. Predictors of Mental Health Crises Among Individuals With Intellectual and Developmental Disabilities Enrolled in the START Program. Psychiatr Serv. 2021 Mar 1;72(3):273-280. doi: 10.1176/appi.ps.202000301. Epub 2020 Dec 18. PMID 33334153
- [Background] Holingue C, Kalb LG, Klein A, Beasley JB. Experiences With the Mental Health Service System of Family Caregivers of Individuals With an Intellectual/Developmental Disability Referred to START. Intellect Dev Disabil. 2020 Oct 1;58(5):379-392. doi: 10.1352/1934-9556-58.5.379. PMID 33032318
- [Background] Kalb LG, Beasley J, Caoili A, Klein A. Improvement in Mental Health Outcomes and Caregiver Service Experiences Associated With the START Program. Am J Intellect Dev Disabil. 2019 Jan;124(1):25-34. doi: 10.1352/1944-7558-124.1.25. PMID 30715923
- [Background] Kalb LG, Beasley J, Klein A, Hinton J, Charlot L. Psychiatric hospitalisation among individuals with intellectual disability referred to the START crisis intervention and prevention program. J Intellect Disabil Res. 2016 Dec;60(12):1153-1164. doi: 10.1111/jir.12330. Epub 2016 Aug 26. PMID 27561378
- [Derived] Kalb LG, Kramer JM, Goode TD, Black SJ, Klick S, Caoili A, Klipsch S, Klein A, Urquilla MP, Beasley JB. Evaluation of telemental health services for people with intellectual and developmental disabilities: protocol for a randomized non-inferiority trial. BMC Health Serv Res. 2023 Jul 25;23(1):795. doi: 10.1186/s12913-023-09663-6. PMID 37491216